CLINICAL TRIAL: NCT03200782
Title: Postprandial Hypoglycemia in Patients After Bariatric Surgery With Empagliflozin and Anakinra - The Hypo-BEAR-Study
Acronym: Hypo-BEAR
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Basel, Switzerland (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Diagnostic
Other Study IDs: EKNZ 2017-00689
Record Dates: First submitted 2017-05-30; First posted 2017-06-27 (Actual); Last update posted 2018-10-24 (Actual); Status verified 2018-10

CONDITIONS: Postprandial Hypoglycemia; Bariatric Surgery; Late Dumping Syndrome
Keywords: postprandial hypoglycemia; bariatric surgery; late dumping syndrome; anakinra; empagliflozin; SGLT2 inhibitor; IL-1Beta; IL1
MeSH Terms: conditions — Hypoglycemia | interventions — empagliflozin; Interleukin 1 Receptor Antagonist Protein; Sodium Chloride

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Placebo-Placebo (Placebo Comparator): subcutaneous placebo (0.67 ml of 0.9% sodium chloride) 3 hours before the test meal and an oral placebo (winthrop tablet) 2 hours before the test meal will be administered by an Independent nurse to the blinded patient
  Interventions: Other: oral placebo (winthrop tablet); Other: subcutaneous placebo (0.67 ml of 0.9% sodium chloride)
- Investigational Drug A Empagliflozin (Active Comparator): subcutaneous placebo (0.67 ml of 0.9% sodium chloride) 3 hours before the test meal and an 10mg of empagliflozin 2 hours before the test meal will be administered by an independent nurse to the blinded patient
  Interventions: Drug: Empagliflozin; Other: subcutaneous placebo (0.67 ml of 0.9% sodium chloride)
- Investigational Drug B Anakinra (Active Comparator): subcutaneous injection of 100mg anakinra 3 hours before the test meal and an oral placebo (winthrop tablet)before the test meal will be administered by an Independent nurse to the blinded patient
  Interventions: Drug: Anakinra; Other: oral placebo (winthrop tablet)

INTERVENTIONS:
Drug: Empagliflozin — Glucose lowering effect of empagliflozin for reducing the counter-regulatory glucose-lowering response
  Arms: Investigational Drug A Empagliflozin
Drug: Anakinra — IL-1Beta blockage effect on insulin secretion and thereby influencing postprandial glucose level
  Arms: Investigational Drug B Anakinra
Other: oral placebo (winthrop tablet) — subcutaneous placebo (0.67 ml of 0.9% sodium chloride) 3 hours before the test meal and an oral placebo (winthrop tablet) 2 hours before the test meal will be administered by an Independent nurse to the blinded patient
  Arms: Investigational Drug B Anakinra; Placebo-Placebo
Other: subcutaneous placebo (0.67 ml of 0.9% sodium chloride) — subcutaneous placebo (0.67 ml of 0.9% sodium chloride) will be administered in arm 'Placebo-Placebo' and arm 'drug: Empagliflozin'
  Arms: Investigational Drug A Empagliflozin; Placebo-Placebo

SUMMARY:
The purpose of the study is to investigate whether hypoglycaemia observed after food intake in bariatric patients can be either influenced by an SGLT2 inhibitor, empagliflozin, or via inhibition of inflammation with an human interleukin-1 receptor antagonist (IL1-RA, anakinra).

DETAILED DESCRIPTION:
Postprandial hypoglycemia also referred as late-dumping after bariatric surgery can be clinically asymptomatic but also life-threatening. The exact mechanisms leading to postprandial hypoglycemia are not fully understood and therapeutic options are limited and often accompanied with reduced life-quality and weight gain.

In this study, prospective, randomly selected and double-blinded treatment is performed to investigate the effect on postprandial hypoglycemia. A total of 12 subjects participate in the study. After a screening date, three study dates will be performed. Participation in the study usually takes two weeks, but can also be extended to three weeks in individual cases. The University Hospital Basel will be the only test center in this study.

In order to check whether the increase in blood glucose after food intake and subsequent excessive reaction of the body followed by hypoglycaemia patients receive either anakinra as a subcutaneous injection 3h or empagliflozin as a tablet 2 h before a liquid standardized test meal. On one study day only subcutaneous and oral placebo control will be used.

At the beginning of each study date as well as at the time of the test meal several blood samples will be taken to evaluate blood glucose and blood glucose-influencing parameters (insulin / C-peptide, intestinal hormones, inflammatory parameters such as C-reactive protein, IL1beta and IL1-receptor agonist as well as macrophage and t-lymphocyte subpopulations) will be controlled. Questionnaires for dumping symptoms (Dumping Rating scale, Sigstad Score) and hypoglycemia testing with mini-mental test, stanford sleepiness scale and Edinburgh Hypoglycemia Scale will be performed repetitively.

ELIGIBILITY:
Inclusion Criteria:

* Patients after roux-y-gastric bypass or biliopancreatic diversion with documented hypoglycemia, i. e. ≤ 2.5 mmol/l and hypoglycaemic symptoms.
* For subjects with reproductive potential, willingness to use contraceptive measures adequate to prevent the subject or the subject's partner from becoming pregnant during the study

Exclusion Criteria:

* Signs of current infection
* Use of any investigational drug in the last four weeks prior to enrolment
* Use of any anti-diabetic drugs
* adrenal insufficiency and/or substitution with glucocorticoids
* Neutropenia (leukocyte count < 1.5 × 109/L or absolute neutrophil count (ANC) < 0.5 × 109/L)
* Anemia (hemoglobin < 11 g/dL for males, < 10 g/dL for females)
* Clinically significant kidney or liver disease (creatinine > 1.5 mg/dL, aspartate aminotransferase (AST)/alanine aminotransferase (ALT) > 2 × ULN, alkaline phosphatase > 2 × ULN, or total bilirubin [tBili] > 1.5 × ULN)
* Current immunosuppressive treatment or documented immunodeficiency
* Uncontrolled congestive heart failure
* Uncontrolled malignant disease
* Currently pregnant or breastfeeding
* known lactose intolerance

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2017-05-30 (Actual); Primary Completion 2018-09-21 (Actual); Study Completion 2018-09-21 (Actual)

PRIMARY OUTCOMES:
Postprandial hypoglycemia in patients after bariatric surgery | 6 hours
  To assess whether empagliflozin or anakinra compared to placebo reduce the severity of hypoglycemia (i.e. change of blood glucose level in mmol/l) following a mixed-meal in patients after bariatric surgery.

SECONDARY OUTCOMES:
change of C-peptide | 6 hours
  plasma level of c-peptide with anakinra or empagliflozin in comparison to placebo
plasma level of IL-1Beta | 6 hours
  plasma level of IL-1Beta with anakinra or empagliflozin in comparison to placebo
plasma level of Glucagon-like Peptide1 (GLP1) | 6 hours
  plasma level of GLP1 with anakinra or empagliflozin in comparison to placebo
change of glucagon level | 6 hours
  plasma level of glucagon with anakinra or empagliflozin in comparison to placebo
changes in Edinburgh Hypoglycemia Scale | 6 hours
  changes in Edinburgh Hypoglycemia Scale with anakinra or empagliflozin in comparison to placebo
amount of glucose needed for restoring normoglycemia | 6 hours
  amount (gramme) of glucose needed for restoring normoglycemia with anakinra or empagliflozin in comparison to placebo
length of time needed for restoring normoglycemia | 6 hours
  length of time (minutes) needed for restoring normoglycemia with anakinra or empagliflozin in comparison to placebo

CONTACTS AND LOCATIONS:
Overall Officials: Marc Donath, MD, Prof., Principal Investigator — University Hopsital Basel
Locations (1):
- University Hospital Basel, Department of Endocrinology, Diabetes and Metabolism, Basel, Switzerland

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Hepprich M, Wiedemann SJ, Schelker BL, Trinh B, Starkle A, Geigges M, Loliger J, Boni-Schnetzler M, Rudofsky G, Donath MY. Postprandial Hypoglycemia in Patients after Gastric Bypass Surgery Is Mediated by Glucose-Induced IL-1beta. Cell Metab. 2020 Apr 7;31(4):699-709.e5. doi: 10.1016/j.cmet.2020.02.013. Epub 2020 Mar 19. PMID 32197070